CLINICAL TRIAL: NCT01998516
Title: Emotional Intelligence in Schizophrenia and Bipolar I Disorder: a Comparison Between Patients, Their Siblings, and Healthy Controls
Brief Title: Emotional Intelligence in Schizophrenia and Bipolar-I- Disorder
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Collaborators: Paracelsus Medical University (Other); Austrian Science Fund (FWF) (Other)
Responsible Party: Principal Investigator, Assoc. Prof. Dr. Alex Hofer, Assoc. Prof. Dr., Medical University Innsbruck
Other Study IDs: KLI 366
Record Dates: First submitted 2013-11-12; First posted 2013-11-29 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Schizophrenia; Bipolar I Disorder
Keywords: Emotional Intelligence
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Schizophrenia Patients
- Bipolar I Patients
- Siblings of Schizophrenia Patients
- Siblings of Bipolar I Patients
- Healthy Controls

SUMMARY:
Scientific Background

Emotional Intelligence (EI) as a part of social cognition is a rather new area of interest which focuses on personality traits and abilities enabling people to cope with both their own feelings as well as those of others. The "Mayer-Salovey-Caruso-Emotional-Intelligence-Test" (MSCEIT) (1) represents a valid and reliable instrument which exclusively covers the emotional components of social cognition. Recent findings indicate, that social cognitive impairments are useful vulnerability indicators and that EI could be an endophenotype for schizophrenia and bipolar I disorder (BD I). To confirm the endophenotype theory, studies concerning EI in relatives of schizophrenia and bipolar patients are needed. To date, studies on EI in BD patients as well as in first degree relatives of patients with schizophrenia or BD haven't been conducted yet. Accordingly, the current study focuses on the four categories assessed by the MSCEIT and aims to compare the task performance of patients, their first degree relatives and healthy control subjects. We assume that the task performance of relatives lies between that of patients and controls. The confirmation of this assumption would verify the trait marker hypothesis and could be a next step to identify a heritable endophenotype for schizophrenia and BD.

Hypotheses

Compared to healthy control subjects patients suffering from schizophrenia or BD I show deficits in EI. Siblings of patients with schizophrenia or BD I show deficits in EI and their task performance lies between that of patients and healthy controls. Deficits in EI are more pronounced in schizophrenia patients than in patients with BD I and are more pronounced in siblings of schizophrenia patients than in siblings of patients with BD I. Independently of diagnosis, deficits in EI affect patients' functional and subjective outcomes.

Methods

Emotional Intelligence will be examined using the MSCEIT in patients with schizophrenia, siblings of schizophrenia patients, patients with BD I, siblings of BD I patients and healthy volunteers matched for age, sex, and educational level. Structured clinical interviews according to DSM-IV (M.I.N.I. + SCID II) will be carried out to assure the diagnosis of schizophrenia or bipolar disorder as well as to detect (comorbid) Axis I and Axis II psychiatric disorders (patients, siblings, control subjects). Functional outcome will be assessed by using the GAF (Global Assessment of Functioning Scale) and the PSP (Personal and Social Performance Scale), subjective quality of life will be examined using the BELP (Berliner Lebensqualiätsprofil). The MWT-B (Multiple choice vocabulary test) will be used to assess premorbid intelligence.

ELIGIBILITY:
Inclusion Criteria:

* ICD-10 diagnosis of schizophrenia or BD (verified by Mini International Neuropsychiatric Interview (M.I.N.I.)
* Outpatients with stable psychopathology for at least half a year and fixed treatment regimen for at least one month prior to testing
* Age: 18-65 years
* Native German Speakers
* Written informed consent

Exclusion Criteria:

* Other axis 1 disorder (verified by M.I.N.I.)
* History of organic mental disorder
* Mental Retardation
* Epilepsy
* Pregnancy/breast-feeding
* Unstable and/or severe organ system diseases, e.g. cardiovascular, endocrine, metabolic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Psychiatric out- and inpatient setting
Sampling Method: Non-Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Emotional Intelligence | 24 month
  Assessed with the MSCEIT (Mayer-Salovey-Caruso-Emotional-Intelligence-Test

SECONDARY OUTCOMES:
Quality of Life | 24 month
  Assessed with the Lancashire Quality of Life Profile

CONTACTS AND LOCATIONS:
Overall Officials: Alex Hofer, Assoc. Prof. Dr., Principal Investigator — Medical University Innsbruck
Locations (1):
- Medical University Innsbruck, Innsbruck, Austria